CLINICAL TRIAL: NCT05815004
Title: Guard3: An Open-label, Parallel-arm, Randomized, Controlled, Phase 2/Phase 3 Study Evaluating the Efficacy and Safety of Autologous HSC Gene Therapy, AVR-RD-02, Compared to ERT for Gaucher Disease Type 3 in Participants Aged 2 to 25
Brief Title: An Efficacy and Safety Study of AVR-RD-02 Compared to Enzyme Replacement Therapy for Treatment of Gaucher Disease Type 3
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Further development of programs halted
Sponsor: AVROBIO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVRO-RD-02-301
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Gaucher Disease, Type 3
Keywords: Gaucher Disease; Gaucher Disease, Type 3; Neuronopathic Gaucher Disease; GD3
MeSH Terms: conditions — Gaucher Disease | interventions — Genetic Therapy; imiglucerase; Velaglucerase alfa, human; taliglucerase alfa

STUDY DESIGN:
Intervention Model Description: Participants, who are randomized to the ERT control arm, will have the opportunity to cross over and receive AVR-RD-02 gene therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVR-RD-02 Arm (Experimental): Participants will have been on a stable prescribed ERT dose for at least 6 consecutive months at the time of Screening and willing to remain on the same ERT dose until 2 weeks prior to gene therapy infusion.
  Interventions: Drug: Gene therapy
- ERT Control Arm (Active Comparator): Participants on stable prescribed ERT dose for at least 6 consecutive months at the time of Screening.
  Participants will have the opportunity to receive a gene therapy infusion of AVR-RD-02 after week 52 of Part 1.
  Interventions: Drug: Gene therapy; Drug: Enzyme Replacement Agent

INTERVENTIONS:
Drug: Gene therapy — AVR-RD-02 Drug product: active substance is autologous CD34+ enriched hematopoietic stem cells (HSCs) that have been genetically modified ex vivo with a lentiviral vector (LV) to contain a ribonucleic acid (RNA) transcript that, after reverse transcription, results in codon-optimized, complementary deoxyribonucleic acid (cDNA) that, upon its integration into human genome, encodes for functional human glucocerebrosidase (GCase)
  Other Names: AVR-RD-02
Drug: Enzyme Replacement Agent — A hydrolytic lysosomal glucocerebrosidase-specific enzyme
  Other Names: Imiglucerase; velaglucerase; taliglucerase alfa
  Arms: ERT Control Arm

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of autologous hemotopoietic stem cell (HSC) gene therapy, AVR-RD-02, compared to enzyme replacement therapy, for the treatment of Gaucher disease Type 3 in male and female participants aged 2 to 25 years.

The study will consist of 2 parts - Core (Part 1) followed by the ERT-crossover (Part 2)

DETAILED DESCRIPTION:
Core (Part 1)

Once a participant consents, he/she will complete the screening period within 30 days.

Eligible participants will have baseline assessments completed 30 days later and then will be randomized into one of two treatment arms: AVR-RD-02 arm or ERT control arm.

If randomized to the AVR-RD-02 arm, the participant will enter the pre-gene therapy infusion period (approximately 15 weeks), which consists of mobilization, apheresis, AVR-RD-02 preparation and testing for release, discontinuation of ERT, and conditioning. The participant will then receive the AVR-RD-02 gene therapy (1 day) followed by a 52-week follow-up period in which periodic safety and efficacy assessments will be performed. Participants will not receive ERT after gene therapy infusion unless indicated by pre-specified laboratory and clinical criteria.

If randomized to the ERT Control arm, the participant will remain on their prescribed ERT regimen for 52-week observation period with approximately 4 study visits during this time.

ERT-crossover (Part 2)

After 52 weeks of observation in Part 1, participants in the ERT Control Arm will have the opportunity to enter Part 2 and receive AVR-RD-02. They will start with baseline assessments and follow a similar schedule to the schedule followed by participants assigned to AVR-RD-02 in the Core Study (Part 1).

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent, caregiver, or legal representative must be willing and able to provide written informed consent/assent for the study in accordance with applicable regulations and guidelines and to comply with all study visits and procedures, including the use of any data collection device(s) that may be used to directly record participant data.
2. Participant is ≥2 to ≤ 25 years old, at the time of providing informed consent or assent.
3. Participant has a confirmed diagnosis of Gaucher disease Type 3 based on all of the following:

   1. Biallelic GBA1 gene mutation
   2. Deficient GCase enzyme activity in blood
   3. Clinical phenotype with the presence of gaze palsy, predominantly horizontal and with slow or absent saccades
4. Participant has the presence of one or both of the following within 3 months of screening:

   1. Ataxia (score ≥1) based on the modified scale for the assessment and rating of ataxia total score (mSARA)
   2. Interstitial lung disease (to be confirmed by radiological imaging)
5. Participant has the presence of one or both of the following within 3 months of screening:

   1. Hepatomegaly
   2. Splenomegaly
6. Participant is on stable prescribed ERT dose for ≥6 consecutive months at the time of Screening.
7. Participant has not received SRT or chaperone therapy for Gaucher disease during the 6 months immediately preceding Screening.
8. Participant is willing to attend all study visits and comply with all study procedures and assessments.
9. Participant is willing to comply with the contraceptive and reproductive requirements.
10. Male and female participants must agree to refrain from donating sperm and eggs, respectively, after undergoing conditioning.
11. Participant must be willing to refrain from donating blood, organs, tissues, or cells for gene therapy infusion any time after AVR-RD-02 treatment.
12. Participant must be willing to receive blood or blood products transfusion to manage AEs as required.

Exclusion Criteria:

1. Participant has a diagnosis of Gaucher disease Type 1 or Type 2.
2. Participant has any one of the following:

   1. Hemoglobin value of <9.0 g/dL
   2. Platelet count of <70 × 109/L
   3. Pulmonary hypertension
   4. Bone crisis attributable to osteonecrosis and/or pathological fractures within 3 months prior to Screening
   5. Treatment refractory epilepsy
   6. Progressive myoclonic epilepsy
3. Participant has had or is scheduled to undergo a partial or total splenectomy.
4. Participant requires use of invasive ventilatory support.
5. Participant requires use of noninvasive ventilator support while awake for longer than 12 hours daily.
6. Participant has a contraindication to ERT, including a prior anaphylactic or anaphylactoid reaction of any severity to ERT.
7. Busulfan is contraindicated for the participant.
8. Participant has a history of sensitivity to dimethyl sulfoxide.
9. Participant presents with iron, folic acid, and/or vitamin B12 deficiency anemia during Screening.
10. Participant has idiopathic thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), thrombocytopenia, anemia, hepatomegaly, splenomegaly, and/or osteoporosis, unrelated to Gaucher disease.
11. Participant has a clinical comorbidity, such as neurologic, cardiovascular, pulmonary, hepatic, gastrointestinal, renal, hematologic, endocrine, metabolic, genetic, immunologic, neoplastic, or psychiatric disease, other medical condition(s), or intercurrent illnesses that may confound the study results or may preclude participation in the study.
12. Participant has a prior or current history of cancer. The one exception is a history of resected squamous cell carcinoma.
13. Participant has any other medical condition that predisposes him/her to (or conveys increased risk of) malignancy, in the opinion of the Investigator.
14. Participant has undergone, or is scheduled to undergo, bone marrow, HSC, and/or solid organ transplant.

    NOTE: Participants who are otherwise eligible for the study but are scheduled for bone marrow transplant or HSC infusion to treat Gaucher disease Type 3 may be enrolled in the study (instead of receiving an allogeneic transplant) and undergo autologous HSC gene therapy with AVR-RD-02.
15. Participant has clinically significant immunosuppressive disease or condition at Screening.
16. Participant is on (or requires treatment with) cytotoxic or immunosuppressive agents from 60 days prior to signing informed consent at Screening (i.e., study enrollment) through the Week 52 study visit; the one exception is treatment with agents required per protocol for autologous HSC infusion.
17. Participant is on (or requires treatment with) red blood cell growth factor (e.g., erythropoietin) from 6 months prior to enrollment (i.e., signing of informed consent at Screening) through the Week 52 study visit.
18. Participant has any condition that makes it impossible to perform magnetic resonance imaging (MRI) studies (including allergies to anesthetics or contrast agents).
19. Participant has medical conditions(s) and/or is receiving medication(s) that would contraindicate ability to undergo mobilization (including contraindication to granulocyte colony stimulating factor [G-CSF] and/or plerixafor), apheresis, or conditioning.
20. Participant has previously received treatment with AVR-RD-02 or any other gene therapy.
21. Participation in (or plan to participate in) any other investigational drug study or plan to be exposed to any other investigational agent, device, and/or procedure from 30 days prior to enrollment (i.e., signing of informed consent at Screening) through study completion.
22. Participant is not suitable for participation as judged by the Investigator, for any reason, including medical or clinical conditions or potential risk of noncompliance to study procedures.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in a multidomain endpoint as assessed by Global Statistical Test (GST) | Baseline to 52 weeks post AVR-RD-02 infusion (AVR-RD-02 arm) or Baseline to 52 weeks (ERT arm)
  The multidomain endpoint consists of the following 4 domains:
  I. Change in modified Scale for Assessment and Rating of Ataxia total score (mSARA)
  II. Percent change in diffusing capacity of the lung for carbon monoxide (DLco) for the assessment of interstitial lung disease (ILD)
  III. Percent change in spleen volume by Magnetic Resonance Imaging (MRI)
  IV. Percent change in a liver volume by MRI

SECONDARY OUTCOMES:
Change from Baseline in Lyso-Gb1 level in cerebrospinal fluid (CSF) as assessed by liquid chromatography tandem mass spectrometry (LC/MS/MS) | Baseline to 52 weeks post AVR-RD-02 infusion (AVR-RD-02 arm) or Baseline to 52 weeks (ERT arm)
Change from baseline in clinical improvement as assessed by Clinical Global Impression -Improvement (CGI-I scale) | Baseline to 52 weeks post AVR-RD-02 infusion (AVR-RD-02 arm) or Baseline to 52 weeks (ERT arm)
Change from baseline in pain as assessed by Brief Pain Inventory-Short Form (BPI-SF) questionnaire scores | Baseline to 52 weeks post AVR-RD-02 infusion (AVR-RD-02 arm) or Baseline to 52 weeks (ERT arm)
Vector Copy Number (VCN) - Engraftment of genetically-modified hematopoietic stem cells (HSCs) in peripheral blood leukocytes (PBL) as assessed by droplet digital polymerase chain reaction (ddPCR) | Baseline to 52 weeks post AVR-RD-02 infusion
Vector Copy Number (VCN) - Engraftment of genetically-modified hematopoietic stem cells (HSCs) in bone marrow as assessed by digital droplet polymerase chain reaction (ddPCR) | Baseline to 52 weeks post AVR-RD-02 infusion
Incidence of clinically significant AEs and SAEs | Baseline to 52 weeks post AVR-RD-02 infusion
Number of participants with clinically relevant abnormalities as assessed by clinical laboratory tests | Baseline to 52 weeks post AVR-RD-02 infusion
Number of participants with clinically relevant abnormalities as assessed by vital signs | Baseline to 52 weeks post AVR-RD-02 infusion
Number of participants with clinically relevant abnormalities as assessed by electrocardiograms (ECGs) | Baseline to 52 weeks post AVR-RD-02 infusion
Number of participants with clinically relevant abnormalities as assessed by physical examinations findings | Baseline to 52 weeks post AVR-RD-02 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Milena Veselinovic, MD, PhD, Study Director — AVROBIO, Inc.

IPD SHARING:
Plan to Share IPD: Yes